CLINICAL TRIAL: NCT07239583
Title: A Description of the Proportion, Genotype Distribution of Respiratory Syncytial Virus and the Severity of Disease in Hospitalized Elderly in Vietnam
Brief Title: Genotype and Disease Burden of RSV in Older Vietnamese Adults (RSV: Respiratory Syncytial Virus )
Acronym: RSV-VN-Elderly
Status: Recruiting | Type: Observational
Sponsor: Tam Anh Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: TA-0003
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Syncytial Virus Infection; Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus (RSV); Acute Respiratory Infection (ARI); Metagenomic Sequencing (mNGS); RSV Genotype; Disease Severity; Healthcare Resource Utilization
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal and sputum samples stored at -70°C for viral PCR and metagenomic sequencing; no human DNA extracted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational, prospective, multicenter study aims to estimate the proportion of RSV infection in adults aged 60 years and older hospitalized due to acute respiratory infections or exacerbation of cardiopulmonary disease.

DETAILED DESCRIPTION:
This is an observational, prospective, multicenter study will enroll 1000 adult patients at Tam Anh TP. Ho Chi Minh General Hospital and Tam Anh General Hospital. The primary outcome is to estimate the proportion of RSV infection in adults aged 60 years and older hospitalized due to acute respiratory infections or exacerbation of cardiopulmonary disease. The secondary outcomes include RSV genotype distribution, viral load, prevalence of co-infections (influenza and COVID-19), clinical and laboratory characteristics associated with disease severity, and patterns of healthcare resource use during and after hospitalization. Analyses will be descriptive. Comparisons between RSV and non-RSV cases will use chi-square or Fisher's exact tests for categorical variables and t-tests or Wilcoxon tests for continuous variables. Logistic regression and Bayesian Model Averaging (BMA) will explore predictors of severe RSV infection.

Eligible patients (≥60 years old) admitted with ARI or acute exacerbations of chronic cardiopulmonary disease will be consecutively screened and enrolled after written informed consent. The study is non-interventional; all participants will receive standard of care treatment at the study sites. Screening will be performed using hospital databases, and medical records will be reviewed to confirm inclusion and exclusion criteria. Demographic, clinical, and epidemiological data will be collected through direct interviews and medical record review.

Within 24 hours of consent, nasopharyngeal swabs (and sputum for patients with lower respiratory symptoms) will be collected by trained nurses. Samples will be placed in viral transport medium, transported to the Clinical Laboratory Center at 2-8°C within 4 hours, and stored at -70°C until testing. All samples will be tested for RSV (A/B), influenza A and B, and SARS-CoV-2 using qualitative PCR. For RSV-positive cases, droplet digital PCR (ddPCR) will quantify viral load. A subset of 200 samples (mNGS subset) will undergo metagenomic next-generation sequencing (mNGS) to determine RSV genotypes and identify other respiratory pathogens. The subset will be selected using an Outcome Dependent Sampling (ODS) method based on disease severity.

During hospitalization, data will be collected on clinical presentation, laboratory and imaging results, comorbidities, treatment course, and outcomes. Disease severity will be assessed using the Respiratory Infection Intensity and Impact Questionnaire (RiiQ™) and CURB-65 score at admission. Treatment information (medications, respiratory support, ICU admission, renal replacement therapy, ECMO, hospital stay duration, and mortality) will be recorded.

A three-month post-discharge follow-up via telephone will evaluate health status and healthcare resource utilization. Data will include readmissions, ICU admissions, outpatient visits, diagnostic tests, and medication use. Investigators will attempt up to three contact calls to reach each participant or caregiver.

All study procedures follow Good Clinical Practice (GCP) and the Declaration of Helsinki. Ethical approval will be obtained from Institutional Review Boards before initiation. Written informed consent will be required. Participant data will be de-identified and securely stored with restricted access. Only trained and authorized staff will handle samples and data.

This study will be the first multicenter prospective investigation of RSV burden and genotypes in older adults in Vietnam. Results will provide baseline epidemiologic data, improve understanding of RSV-related hospitalization in the elderly, and inform prevention and vaccination strategies. The use of ddPCR and mNGS will generate high-resolution data on viral load, pathogen co-detection, and genomic diversity, contributing to the global understanding of RSV epidemiology and supporting future RSV vaccine policy development in Vietnam.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in the study, participants must meet all inclusion criteria:

1. Individuals ≥ 60 years old at the time of screening (calculated from the date of birth to the date of screening)
2. ARI or exacerbation of cardiopulmonary diseases diagnosed at the time of admission. ARI or ARI-compatible symptoms were defined as either:

   * New onset or increase from baseline of: nasal congestion, rhinorrhea, sore throat, hoarseness, cough, sputum production, dyspnea, wheezing, hypoxemia, or
   * Admitting diagnosis suggestive of ARI (e.g., pneumonia, upper respiratory infection, bronchitis, influenza, cough, viral respiratory illness, respiratory distress, or respiratory failure), or
   * Admitting diagnosis was the exacerbation of an underlying cardiac or pulmonary disease involving acute respiratory symptoms within the previous 2 weeks (e.g., congestive heart failure [CHF], chronic obstructive pulmonary disease [COPD], or asthma exacerbation).
3. The participant agrees to voluntarily participate in this study.

Exclusion Criteria:

To be enrolled in the study, participants must have none of the exclusion criteria:

1. Symptom onset > 6 days prior to screening date
2. Acute symptoms confirmed to be unrelated to infection or as assessed by the investigator
3. Admission to any hospital within the 30 days preceding the screening date
4. Previously enrolled in the study in the last 45 days

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adults aged ≥60 years with acute respiratory infections at Tam Anh TP. Ho Chi Minh General Hospital and Tam Anh General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of RSV infection in adults aged 60 years and older hospitalized due to acute respiratory infections or exacerbation of cardiopulmonary disease. | Within 24 hours after hospital admission
  The proportion of participants with laboratory-confirmed RSV infection (including RSV A and RSV B) among adults aged ≥60 years hospitalized for acute respiratory infection or cardiopulmonary disease exacerbation. Diagnosis will be based on qualitative PCR results from nasopharyngeal or sputum samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Tam Anh TP. Ho Chi Minh General Hospital, Ho Chi Minh City, Southern Vietnam, Vietnam

IPD SHARING:
Plan to Share IPD: No